CLINICAL TRIAL: NCT03810469
Title: Perfusion Analysis of the Foot in Patients With Critical Limb Ischemia Before and After Revascularization and Predictive Value on Amputation-free Survival
Brief Title: Foot Perfusion Analysis to Predict Limb Salvage
Acronym: DELTA-PERF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier de Valenciennes (Network)
Responsible Party: Sponsor
Other Study IDs: 2018-01
Record Dates: First submitted 2019-01-15; First posted 2019-01-18 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Critical Limb Ischemia; Peripheral Arterial Disease
Keywords: limb salvage; foot perfusion; hybrid room
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at evaluating the correlation between foot perfusion on angiographies performed before and after revascularization and limb salvage in patients with critical limb ischemia.

DETAILED DESCRIPTION:
Critical limb ischemia (CLI) in diabetic patients is increasing drastically worldwide, and is already recognized as a major health issue. CLI is frequently leading to major amputations. Therefore, one of the key point to prevent limb loss is to restore a good vascularization to the foot, usually thanks to endovascular means.

No consensual indicator is currently available to estimate if the limb revascularization will be sufficient or not to prevent amputation, and to help physicians decide if they should be more aggressive during the endovascular procedure. Transcutaneous oximetry and value of the ankle-brachial index (ABI) are commonly used in the ward (not available in the operating room), but have shown poor correlation to wound healing or limb salvage and results are frequently biased because of the arterial wall calcifications due to diabetes. Value of the first toe systolic pressure is currently under evaluation to predict survival without amputation, with promising results, but cannot be applied to patients with wounds at this level or previous minor amputation.

The emergence of hybrid rooms in the operating theater offer access to high quality imaging and image post-treatment. Those capabilities could be used to analyze the flow and the tissue perfusion in the foot, and correlate those imaging parameters to positive clinical outcomes, such as wound healing, thus creating a useful tool to guide physicians in daily practice.

Differences between foot angiographies performed before and after revascularization could be used to estimate the quality of the revascularization and predict wound healing and limb salvage. This method would be directly available in the operating room and could help physicians to optimize their strategy during the procedure

ELIGIBILITY:
Inclusion Criteria:

* Patients with critical limb ischemia Rutherford 4, 5 and 6, with at least one pre-operative exam (CTA, magnetic resonance angiography or ultrasound) demonstrating a peripheral arterial disease, and requiring an endovascular or hybrid (meaning combined with a surgical technique) revascularization of the lower limb.

Exclusion Criteria:

* Patients not willing to give their consent to study enrollment
* Patients under 18 years old
* Patients with severe renal insufficiency (estimated creatinine clearance < 30 mL/min), without dialysis
* Patients with life threatening septic wounds who would require an amputation at the initial presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from peripheral arterial disease in critical limb ischemia (Rutherford 4, 5 and 6) at the initial presentation, with a major risk of limb amputation at mid-term without revascularization.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-10-02 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with major amputation | 1 month
  Major amputations are defined as below or above the knee amputations on the treated limb. This is a clinical binary criterion (0=Freedom from major amputation, 1=Major amputation)
Number of participants with major amputation | 3 months
  Major amputations are defined as below or above the knee amputations on the treated limb. This is a clinical binary criterion (0=Freedom from major amputation, 1=Major amputation)
Number of participants with major amputation | 6 months
  Major amputations are defined as below or above the knee amputations on the treated limb. This is a clinical binary criterion (0=Freedom from major amputation, 1=Major amputation)
Number of participants with major amputation | 1 year
  Major amputations are defined as below or above the knee amputations on the treated limb. This is a clinical binary criterion (0=Freedom from major amputation, 1=Major amputation)

SECONDARY OUTCOMES:
Wound Healing | 1 month
  Complete wound Healing at the level of the foot according to the WiFI classification
Wound Healing | 3 months
  Complete wound Healing at the level of the foot according to the WiFI classification
Wound Healing | 6 months
  Complete wound Healing at the level of the foot according to the WiFI classification
Wound Healing | 1 year
  Complete wound Healing at the level of the foot according to the WiFI classification
Number of patients with secondary intervention | 1 year
  Number of participants with a secondary intervention. Secondary intervention is defined as all secondary surgical interventions (both endovascular and open repairs) associated to critical limb ischemia on the same limb. It includes secondary angioplasties, bypasses or minor and major amputations. This is a clinical binary criterion (0= Freedom from secondary intervention, 1=At least one secondary intervention)
Overall Mortality | 1 year
  Overall Mortality, all-cause included

CONTACTS AND LOCATIONS:
Locations (1):
- CH Valenciennes, Valenciennes, France

REFERENCES:
- [Result] Brownrigg JR, Apelqvist J, Bakker K, Schaper NC, Hinchliffe RJ. Evidence-based management of PAD & the diabetic foot. Eur J Vasc Endovasc Surg. 2013 Jun;45(6):673-81. doi: 10.1016/j.ejvs.2013.02.014. Epub 2013 Mar 27. PMID 23540807
- [Result] Wang Z, Hasan R, Firwana B, Elraiyah T, Tsapas A, Prokop L, Mills JL Sr, Murad MH. A systematic review and meta-analysis of tests to predict wound healing in diabetic foot. J Vasc Surg. 2016 Feb;63(2 Suppl):29S-36S.e1-2. doi: 10.1016/j.jvs.2015.10.004. PMID 26804365
- [Result] Wickstrom JE, Laivuori M, Aro E, Sund RT, Hautero O, Venermo M, Jalkanen J, Hakovirta H. Toe Pressure and Toe Brachial Index are Predictive of Cardiovascular Mortality, Overall Mortality, and Amputation Free Survival in Patients with Peripheral Artery Disease. Eur J Vasc Endovasc Surg. 2017 May;53(5):696-703. doi: 10.1016/j.ejvs.2017.02.012. Epub 2017 Mar 11. PMID 28292565
- [Result] Brownrigg JR, Hinchliffe RJ, Apelqvist J, Boyko EJ, Fitridge R, Mills JL, Reekers J, Shearman CP, Zierler RE, Schaper NC; International Working Group on the Diabetic Foot. Performance of prognostic markers in the prediction of wound healing or amputation among patients with foot ulcers in diabetes: a systematic review. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:128-35. doi: 10.1002/dmrr.2704. PMID 26342129